CLINICAL TRIAL: NCT01247207
Title: An Open-Label, Safety Study for Ataluren (PTC124) Patients With Nonsense Mutation Dystrophinopathy
Brief Title: Study of Ataluren in Previously Treated Participants With Nonsense Mutation Dystrophinopathy (nmDBMD)
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC124-GD-016 DMD
Record Dates: First submitted 2010-11-22; First posted 2010-11-24 (Estimated); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne muscular dystrophy; Becker muscular dystrophy; Nonsense mutation; Premature stop codon; DMD; BMD; nmDBMD; DBMD; Ataluren; PTC124
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — ataluren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ataluren (Experimental): Participants will receive 3 doses of ataluren oral suspension per day (10 mg/kg in the morning, 10 mg/kg at mid-day and 20 mg/kg in the evening).
  Interventions: Drug: Ataluren

INTERVENTIONS:
Drug: Ataluren — Ataluren will be administered as per the dose and schedule specified in the arm.
  Other Names: PTC124; Translarna

SUMMARY:
The objective of this study is to assess the safety and tolerability of 10, 10, 20 milligrams per kilogram (mg/kg) ataluren in participants with nmDBMD who had prior exposure to ataluren in a PTC sponsored clinical trial or treatment plan, and siblings of those participants (provided those participants have completed the placebo-controlled portion of the trial).

The treatment will continue under this protocol until consent withdrawal by participants, withdrawal due to worsen condition after initiating ataluren treatment, withdrawal by investigator, withdrawal due to participant unable to tolerate ataluren, participant is eligible to participate in another ataluren nmDBMD clinical trial program initiated by sponsor, study is discontinued by the relevant regulatory authority and/or sponsor, or until ataluren becomes commercially available.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of signed and dated informed consent/assent document(s) indicating that the participant (and/or his parent/legal guardian) has been informed of all pertinent aspects of the trial. Note: If the study candidate is considered a child under local regulation, a parent or legal guardian must provide written consent prior to initiation of study screening procedures and the study candidate may be required to provide written assent. The rules of the responsible Institutional Review Board/Independent Ethic Committee (IRB/IEC) regarding whether one or both parents must provide consent and the appropriate ages for obtaining consent and assent from the participant should be followed.
* History of exposure to ataluren in a prior PTC study or treatment plan and effected nmDBMD siblings of those participants (provided those participants have completed the placebo-controlled portion of the trial).
* Fertile men, who are sexually active with women of childbearing potential and who have not had a vasectomy, must agree to use a barrier method of birth control during the study and for up to 50 days after the last dose of study drug.
* Willingness and ability to comply with scheduled visits, drug administration and return plan, study procedures, laboratory tests, and study restrictions Note: Psychological, social, familial, or geographical factors that might preclude adequate study participation should be considered.

Exclusion Criteria:

* Exposure to another investigational drug within 1 month prior to start of study treatment.
* Eligibility for another ataluren clinical trial that is actively enrolling study participants.
* Positive for Hepatitis B core antibody or Hepatitis C antibody at screening for ataluren naïve participants (siblings) or participants who have a temporary treatment gap of 1 year before entering study
* Known hypersensitivity to any of the ingredients or excipients of ataluren (refined polydextrose, polyethylene glycol 3350, poloxamer 407, mannitol 25C, crospovidone XL10, hydroxyethyl cellulose, colloidal silica, magnesium stearate).
* Ongoing intravenous (IV) aminoglycoside or IV vancomycin therapy.
* Ongoing uncontrolled medical/surgical condition, electrocardiogram (ECG) findings, or laboratory abnormality that, in the investigator's opinion, could adversely affect the safety of the participant or make it unlikely that follow-up would be completed.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2010-11-30 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events | Baseline up to end of study (up to approximately 8 years)
Number of Participants With Laboratory Parameters Abnormalities | Baseline up to end of study (up to approximately 8 years)
  Laboratory parameters include hematological, serum biochemistry, adrenal laboratories, and urine data.
Number of Participants With Abnormal Physical Findings | Baseline up to end of study (up to approximately 8 years)
  Physical findings include weight, physical examination data, systolic and diastolic blood pressure, radial pulse rate, and body temperature.

CONTACTS AND LOCATIONS:
Overall Officials: Vinay Penematsa, MD, Study Director — PTC Therapeutics, Inc.
Locations (34):
- United States (29):
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Children's Hospital of Los Angeles, Los Angeles, California
  - UCLA, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of California-Davis, Sacramento, California
  - University of CA, San Francisco-Benioff Children's Hospital, San Francisco, California
  - Children's Hospital Colorado - Center for Cancer and Blood Disorders, Aurora, Colorado
  - Child Neurology Center of NW Florida NW, Gulf Breeze, Florida
  - Rare Disease Research, LLC, Atlanta, Georgia
  - Rush Univ Medical Center, Chicago, Illinois
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Children's Hospital of Boston/Harvard Medical School, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University Medical School, St Louis, Missouri
  - Columbia University Pediatric Neuromuscular Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Shriners Hospital for Children-Portland, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Childrens Medical Center Dallas, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
- Canada (5):
  - Alberta Children's Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - London Health Sciences Centre, London, Ontario
  - Children's Hospital of East Ontario, Ottawa, Ontario
  - CHU de Québec - Université Laval, Québec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hirawat S, Welch EM, Elfring GL, Northcutt VJ, Paushkin S, Hwang S, Leonard EM, Almstead NG, Ju W, Peltz SW, Miller LL. Safety, tolerability, and pharmacokinetics of PTC124, a nonaminoglycoside nonsense mutation suppressor, following single- and multiple-dose administration to healthy male and female adult volunteers. J Clin Pharmacol. 2007 Apr;47(4):430-44. doi: 10.1177/0091270006297140. PMID 17389552
- [Result] Welch EM, Barton ER, Zhuo J, Tomizawa Y, Friesen WJ, Trifillis P, Paushkin S, Patel M, Trotta CR, Hwang S, Wilde RG, Karp G, Takasugi J, Chen G, Jones S, Ren H, Moon YC, Corson D, Turpoff AA, Campbell JA, Conn MM, Khan A, Almstead NG, Hedrick J, Mollin A, Risher N, Weetall M, Yeh S, Branstrom AA, Colacino JM, Babiak J, Ju WD, Hirawat S, Northcutt VJ, Miller LL, Spatrick P, He F, Kawana M, Feng H, Jacobson A, Peltz SW, Sweeney HL. PTC124 targets genetic disorders caused by nonsense mutations. Nature. 2007 May 3;447(7140):87-91. doi: 10.1038/nature05756. Epub 2007 Apr 22. PMID 17450125
- See also: PTC Therapeutics, Inc website — http://www.ptcbio.com
- See also: Protocol V7.0 — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217411&parentIdentifier=PTC124-GD-016%20DMD&attachmentIdentifier=2d0b5df7-f526-4813-bd6c-3fb06c5f83dc&fileName=PTC124-GD-016-DMD_Protocol_V7.0_with_PDMS-2.pdf&versionIdentifier=